CLINICAL TRIAL: NCT06967740
Title: Epidemiological Factors and Optimization of Conservative Approaches to Precancerous Lesions of Female Reproductive Organs
Status: Recruiting | Type: Observational
Sponsor: Nikola Janovska (Other Government)
Responsible Party: Sponsor-Investigator, Nikola Janovska, Medical doctor, Department of Gynecology and Obstetrics, Faculty Hospital Kralovske Vinohrady
Organization: Faculty Hospital Kralovske Vinohrady (Other Government)
Other Study IDs: EKVP/51/2024
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia (CIN); Risk Factors; Conservative Management
Keywords: Cervical Intraepithelial Neoplasia (CIN); Conservative management; Precancerous cervical lesions
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cytology, cervical biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Unvaccinated: Without adjuvant vaccination for HPV
- Vaccinated: Adjuvantly vaccinated against HPV with Gardasil-9

SUMMARY:
The primary aim of this study is to develop a recommended clinical practice guideline for managing women with HPV HR (high-risk human papillomavirus) positivity and cervical lesions. Additionally, in collaboration with the Bioptic Laboratory, the study will analyze the integration of HPV HR testing into screening programs for women aged 35, 45, and 55, with a focus on optimizing management strategies for HPV HR-positive women.

Research Objectives:

* Evaluate spontaneous regression/progression over two years based on HPV HR genotyping (three groups - according to Alinity: high, intermediate, and low risk).
* Assess spontaneous regression/progression over two years based on HPV HR genotyping and viral load in HPV-vaccinated vs. non-vaccinated patients.
* Evaluate spontaneous regression/progression over two years based on methylation results.
* Assess spontaneous regression/progression over two years based on CinTec plus results.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* cervical biopsy - HG lesion
* Age: 18-46 years
* colposcopicaly visible transformation zone
* HPV: Unvaccinated
* cytology all except AIS, adenocarcinoma, squamous cell carcinoma, AGC NEO

Exclusion Criteria:

* cytology AIS, AGC NEO, adenocarcinoma, squamous cell carcinoma
* immunosuppression
* active autoimmune disease
* history of cervical cryodestruction
* HPV vaccinated prior to start of the study

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Females with HG precancerous lesions of the cervix.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate spontaneous regression/progression over a 2-year period according to HPV HR genotyping | 2 year follow up
  Evaluate the risk of regression or progression of cervical lesion in patients with HG (high-grade) cervical precancerous lesion - according to stratification of HPV genotyping
To evaluate spontaneous regression/progression over a 2-year period according to methylation results | 2 year follow up
  Evaluate the risk of regression or progression of cervical lesion in patients with HG cervical precancer - according to methylation test (FAM194A, miR124-2)
o evaluate spontaneous regression/progression over a 2-year period according to CinTec plus | 2 year follow up
  Evaluate the risk of regression or progression of cervical lesion in patients with HG cervical precancer - according to CinTec plus test - mmunohistochemical marker utilizing two proteins - p16 and Ki67

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Rob, Prof., MUDr., Csc., Principal Investigator — University Hospital Kralovske Vinohrady
Locations (1):
- University Hospital Kralovske Vinohrady, Prague, Czechia

REFERENCES:
- [Background] Lee MH, Finlayson SJ, Gukova K, Hanley G, Miller D, Sadownik LA. Outcomes of Conservative Management of High Grade Squamous Intraepithelial Lesions in Young Women. J Low Genit Tract Dis. 2018 Jul;22(3):212-218. doi: 10.1097/LGT.0000000000000399. PMID 29762428
- [Background] Kyrgiou M, Athanasiou A, Paraskevaidi M, Mitra A, Kalliala I, Martin-Hirsch P, Arbyn M, Bennett P, Paraskevaidis E. Adverse obstetric outcomes after local treatment for cervical preinvasive and early invasive disease according to cone depth: systematic review and meta-analysis. BMJ. 2016 Jul 28;354:i3633. doi: 10.1136/bmj.i3633. PMID 27469988
- [Background] Depuydt CE, Jonckheere J, Berth M, Salembier GM, Vereecken AJ, Bogers JJ. Serial type-specific human papillomavirus (HPV) load measurement allows differentiation between regressing cervical lesions and serial virion productive transient infections. Cancer Med. 2015 Aug;4(8):1294-302. doi: 10.1002/cam4.473. Epub 2015 May 20. PMID 25991420